CLINICAL TRIAL: NCT04082247
Title: A Cluster Randomized Controlled Trial Evaluating the Effectiveness of a Healthy Lifestyle Program on Childhood Executive Functions
Brief Title: Healthy Children 2021 Study in Childcare Centers
Acronym: HC2021
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Helena Rafaela Vieira do Rosario, Principal Investigator, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: University of Minho
Record Dates: First submitted 2019-09-03; First posted 2019-09-09 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Family Health; Child Health; Sleep; Child; Executive Function; Pediatric Obesity; Dietary Habits
MeSH Terms: conditions — Pediatric Obesity; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The education and training of early childhood educators (developed by the researchers) and their intervention on children.
  Interventions: Behavioral: The education and training of early childhood educators and their intervention on children
- Control group (No Intervention): Receive the standard care.

INTERVENTIONS:
Behavioral: The education and training of early childhood educators and their intervention on children — A 24-week cluster randomized trial will be developed, with the childcare being the randomization unit. Training sessions will be conducted for all early childhood educators in the intervention group. The control group will receive the Portuguese "standard" education and at the end of the intervention this group will also receive the initial training given to the intervention group, so that they can later also implement the intervention. At the end of the intervention, all early childhood educators and parents/guardians will have access to the intervention outcomes.
  Arms: Experimental group

SUMMARY:
In Portugal, 17.3% of children under 10 years old are overweight and 7.7% are obese. Research has shown the implementation of healthy lifestyle promotion programs and obesity prevention, however "best practices" are far from being defined. Also, the first five years of life are important for the executive functions development, namely memory, inhibition (including self-regulation) and flexibility, which includes creative thinking, thinking "outside of the box", important in problem solving. The importance of social and emotional dimensions, as well as physical health for the development of cognitive health is consensual, as sleep deprivation, low physical activity, unhealthy food may inhibit the proper development of executive functions.

This project aims to evaluate the effectiveness of a healthy lifestyle promotion program on emotional, social and cognitive development and eating habits, sleep and physical activity in children between 12 and 42 months of age.

A cluster randomised trial will be developed and 300 children, from 16 childcare centres will be invited to participate. Half of the childcare centres will be allocated to the control group and the other half to the intervention group. Data collection will occur before randomisation (at baseline) and after intervention. A feasibility study will be undertaken prior to the experimental study, in accordance with internationally accepted procedures.

The investigators intend to implement the concept that the development of executive functions requires the combination of healthy eating, physical activity and sleep.

The project will contribute with evidence-based to the cognitive, social and emotional development in children.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy (with no pre-existing conditions) children aged 12-42 months at baseline.

Exclusion Criteria:

* Children with disability

Ages: 12 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change in cognitive, social and emotional development | 12 months - 42 months
  The Bayley Scales of Infant and Toddler Development - III edition identifies the child's developmental competencies across five major developmental domains; identifies deficits in very young children; and determines the need for further in-depth assessment. Raw scores from the cognitive and social-emotional scale, which does not contain separate subtests, can be converted to a scaled score (M=10, SD=3), which can then additionally be converted to a composite score equivalent (M=100, SD=15). Raw scores for cognitive and motor subtests translate to scaled scores based on 10-day increments up to age 5 months 16 days, at which point norms are based on 1-month intervals (e.g., 5 months 16 days to 6 months 15 days, 35 months 16 days to 36 months 15 days). The normative sample for the social-emotional domain is divided into nine age categories (by months: 0-3, 4-5, 6-9, 10-14, 15-18, 19-24, 25-30, and 31-40). Higher values represent a better performance.
Change in dietary intake | 12 months - 42 months
  The child's eating habits will be collected using the one-day food record, completed by parents or early childhood educators.
Change in 24-h movement | 12 months - 42 months
  Physical activity, sleep and sedentary behavior will be assessed using the Actigraph accelerometer, which will be used for 5 consecutive days (3 days a week and 2 days a weekend).

SECONDARY OUTCOMES:
Sociodemographic profile | 12 months - 42 months
  Families' profile will be assessed using the Graffar scale, adapted to Portugal. This is an international social classification, used as an indicator of the various welfare levels of a social group. It includes 5 criteria: occupation, level of education, sources of family income, housing comfort and appearance of the neighbourhood. The sum of the points obtained in the classification provides a final score that corresponds to social class, according to the following classification: Class I (5-9 points), Class II (10-13 points), Class III (14-17 points), Class IV (18-21 points) and Class V (22-25 points). The higher the score, the better the sociodemographic profile.
Family lifestyles | 12 months - 42 months
  Families' lifestyles will be assessed through the International Physical Activity Questionnaire-short version, which looks at the types of intensity of physical activity and sitting time that people do as part of their daily lives. It's composed by 7 items, open-ended questions surrounding individuals' (parents) last 7-day recall of physical activity.
Change in length and waist circumference | 12 months - 42 months
  Length and waist circumference (cm) will be assessed with no clothes nor shoes using standardised procedures.
Change in weight | 12 months - 42 months
  Weight (kg) will be assessed with no clothes and no shoes, using standardised procedures.
Change in blood pressure (systolic and diastolic) | 12 months - 42 months
  Digitally assessed, using standardized procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Rafaela Rosário, Dr, Principal Investigator — University of Minho
Locations (1):
- University of Minho, Braga, Portugal

REFERENCES:
- [Derived] Duarte A, Martins S, Augusto C, Silva MJ, Lopes L, Santos R, Rosario R. The impact of a health promotion program on toddlers' socio-emotional development: a cluster randomized study. BMC Public Health. 2024 Feb 9;24(1):415. doi: 10.1186/s12889-024-17953-9. PMID 38331822